CLINICAL TRIAL: NCT03260140
Title: DVD Lifestyle Intervention (D-ELITE)
Brief Title: DVD Lifestyle Intervention
Acronym: D-ELITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 15-364; I01HX002113 (NIH)
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: weight loss; lifestyle; diet; exercise; randomized controlled trial
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign participants to one of two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- behavioral lifestyle intervention (Experimental): The investigators will provide participants with the the behavioral lifestyle intervention
  Interventions: Behavioral: behavioral lifestyle intervention
- usual care control (No Intervention): participant in this arm will continue with usual care

INTERVENTIONS:
Behavioral: behavioral lifestyle intervention — The investigators will provide participants with the behavioral lifestyle intervention
  Arms: behavioral lifestyle intervention

SUMMARY:
Most Veterans who receive VA healthcare have obesity (41%) or are classified as overweight (37%), putting them at higher risk for multiple serious chronic health conditions. Providing evidence-based behavioral weight management programs to Veterans with obesity is a priority for the VA National Center for Health Promotion and Disease Prevention (NCP). While the VA NCP's MOVE! program-primarily delivered with in-person group visits-helps Veterans with obesity lose weight, its reach has been limited because of various barriers to care. Some Veterans may do better with a program they can complete from home at their own pace. In this trial, study investigators are examining the effectiveness among Veterans of a previously proven self-directed lifestyle intervention (called DVD Lifestyle Intervention (D-ELITE)) that targets modest, clinically meaningful weight loss over the course of a year using recorded video lessons (DVD or online streaming), written self-study aids, and optional lifestyle coaching. The study will compare participants randomly assigned to receive D-ELITE to those continuing in usual care on weight and self-reported general physical health status, one year after enrollment. Secondary outcomes include weight and general physical health status two years after enrollment; and obesity-related biometric measures (blood pressure and HbA1c) and self-report psychological and behavioral factors such as physical activity and sleep quality, at one- and two-years following enrollment.

Veterans with obesity living in the western US were identified using the VA Corporate Data Warehouse (CDW), recruited to participate via mail and telephone, and randomly assigned to receive the study intervention or usual care alone. The study uses CDW to assess weight change and biometric outcomes. To assess self-report outcomes, participants completed questionnaires, by mail or telephone, at baseline and 12 months after randomization, and are currently completing 24-month follow-up questionnaires. The D-ELITE intervention focuses on gradual lifestyle behavior change aimed at improving eating habits and increasing physical activity. It encourages participants to gradually achieve and maintain a 5-10% loss of baseline body weight and at least 150 minutes of moderate-intensity physical activity, such as brisk walking, each week. The D-ELITE intervention program consists of watching one video, completing corresponding written self-guided learning materials, and tracking food intake and physical activity each week for the first 12 weeks, then working through 10 additional written handouts and continued food and activity tracking for the next nine months. Intervention participants have access to a lifestyle coach, as desired, for the full 12-month intervention period. In addition to patient outcomes, this study will examine the cost of delivering the intervention, information relevant to decision-makers and potential future dissemination. Evidence-based programs like this, which can be delivered remotely and with likely minimal resources required from the VA healthcare system, are greatly needed, especially now as the SARS-CoV-2 pandemic has required VA to rapidly transition to providing more remotely-delivered care.

Impact: The DELITE trial has potential to provide the evidence needed for deciding whether a low-cost, low-technology, self-directed program can be used to expand the treatment of obesity to a population-based level by improving access to obesity treatment regardless of Veteran place of residence.

ELIGIBILITY:
Inclusion Criteria:

* Recent VA primary care measured BMI between 30.0-44.9 kg/m2 (at facility in pacific or mountain time zone)
* Access to DVD player or internet
* Able to participate fully in all study protocol/procedures including informed consent

Exclusion Criteria:

* Inability to speak, read, or understand English
* Recent weight loss interventions including use of prescription weight-loss medications, participation in group or individual weight loss programs provided by trained personnel, bariatric surgery (or plans for during the study period)
* Expected weight loss because of alternate explanations such as from illness
* High variability in weight due to fluctuations in volume status (ascites - liver disease, chronic heart failure)
* Safety and/or adherence concerns due to severe physical or mental health issues, or life expectancy <24 months
* Pregnant, lactating, or planning to become pregnant during the study period;
* Participation in other intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Hoerster, PhD MPH BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoerster KD, Collins MP, Au DH, Lane A, Epler E, McDowell J, Baron AE, Rise P, Plumley R, Nguyen T, Schooler M, Schuttner L, Ma J. Testing a self-directed lifestyle intervention among veterans: The D-ELITE pragmatic clinical trial. Contemp Clin Trials. 2020 Aug;95:106045. doi: 10.1016/j.cct.2020.106045. Epub 2020 May 28. PMID 32473403
- [Derived] Hoerster KD, Hunter-Merrill R, Nguyen T, Rise P, Baron AE, McDowell J, Donovan LM, Gleason E, Lane A, Plumley R, Schooler M, Schuttner L, Collins M, Au DH, Ma J. Effect of a Remotely Delivered Self-directed Behavioral Intervention on Body Weight and Physical Health Status Among Adults With Obesity: The D-ELITE Randomized Clinical Trial. JAMA. 2022 Dec 13;328(22):2230-2241. doi: 10.1001/jama.2022.21177. PMID 36511927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Started | 254 | 257
Completed | 249 | 252
Not Completed | 5 | 5
Not completed — Death | 4 | 1
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control | Total
Number analyzed (Participants) | 254 | 257 | 511
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.17) | 58.1 (13.58) | 57.4 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 112 | 230
  Male | 136 | 145 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 29 | 66
  Not Hispanic or Latino | 217 | 223 | 440
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 24 | 32 | 56
  White | 203 | 206 | 409
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Weights were obtained from the VA electronic health record. For the weight variable, baseline is the weight used to identify Veterans for recruitment to participate.
Time Frame: Weight closest to 12 months from baseline between 9-15 months post-baseline
Population: The investigators report here the unadjusted means at 12 months. The analysis population for adjusted between-group differences includes study participants with a measurement at baseline and/or 12-month follow-up; see Statistical Analysis 1 for those results.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 217 | 212
kilogram (kg) | 99.8 (15.8) | 101.0 (15.0)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average 12-month weight between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.001, Mixed Models Analysis; Difference in average weight at 12 months between control and intervention groups; Mean Difference (Final Values) = -1.93, 97.5% CI 2-sided [-3.24 to -0.61] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

2. Primary Outcome: Short Form (SF)-12 PCS
Description: The SF-12 is a health-related quality of life measure that assesses general physical (PCS) and mental health (MCS) functioning and well-being, with the PCS score serving as co-primary outcome. The investigators scored the SF-12 using QualityMetric's scoring software. PCS scores range from 0-100 with higher scores indicating better general physical health.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 191 | 219
score on a scale | 44.3 (10.7) | 43.2 (9.8)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the 12-month SF-12 PCS between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.388, Mixed Models Analysis; Difference in average SF-12 PCS score at 12 months between control and intervention groups; Mean Difference (Final Values) = 0.69, 97.5% CI 2-sided [-1.11 to 2.49] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

3. Secondary Outcome: International Physical Activity Questionnaire (IPAQ)
Description: 7-item short form of the IPAQ, which evaluates weekly walking, vigorous and moderate-intensity activity. The investigators report here the number of participants engaging in at least 150 minutes of activity per week.
Time Frame: 12 months post baseline
Population: The investigators report here the unadjusted number of participants engaging in at least 150 minutes of activity per week. The analysis population for adjusted between-group differences includes study participants with measurements at both baseline and 12 months; see Statistical Analysis 1 for those results.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 193 | 219
Participants | 149 | 143
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Group-specific McNemar's Chi-Square tests were applied to examine the change from baseline to follow-up in dichotomized IPAQ (>=150 vs <150) minutes of physical activity per week. To compare intervention vs. control at 12 months, we applied an F test. The intervention effect was an odds ratio of the ratios of discordant pairs in the intervention vs the control group; Test type: Superiority; p = 0.308, F test-ratio of 2 McNemar's Chi-Squares; Sign test = 1.76, 95% CI 2-sided [0.85 to 3.66]

4. Secondary Outcome: "Starting the Conversation"
Description: 8-item self-report measure of diet quality that assesses intake of various types of food (e.g., fruit and vegetable, sugary beverages). Scores range from 0-16 with higher scores indicating better diet quality.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 191 | 217
score on a scale | 6.2 (2.6) | 6.4 (2.7)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average 12-month score between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.396, Mixed Models Analysis; Difference in average weight at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.61 to 0.24] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Survey Change
Description: 4-item self-report scale indicating sleep disturbance. Raw scores are converted into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher scores represent more sleep disturbance.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 192 | 219
T-score | 52.5 (9.2) | 52.0 (9.3)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.657, Mixed Models Analysis; Difference in average score at 12 months between control and intervention groups; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-1.02 to 1.61] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Related Impairment Survey Change
Description: 8-item self-report scale indicating sleep impairment. Raw scores are converted into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher scores represent more sleep impairment.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 193 | 218
T-score | 51.7 (10.7) | 52.2 (10.3)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.281, Mixed Models Analysis; Difference in average score at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.33 to 0.68] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

7. Secondary Outcome: Dietary Self-efficacy
Description: Three items measuring diet self-efficacy from the Patient-centered Assessment and Counseling for Exercise plus Nutrition (PACE+) Adult Psychosocial Questionnaire. Scores range from 1-5 with higher scores representing higher diet self-efficacy.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 193 | 219
score on a scale | 3.1 (1.0) | 3.0 (1.0)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average score between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.483, Mixed Models Analysis; Difference in average score at 12 months between control and intervention groups; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.11 to 0.23] — Standard errors estimated using Kenward-Rodgers adjustment for the denominator degrees of freedom

8. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: HbA1c values were obtained from the VA electronic health record. HbA1c is a measure of the percentage of glucose in the blood.
Time Frame: HbA1c closest to 12 months from baseline between 9-15 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 135 | 133
percentage of glycosylated hemoglobin | 6.3 (1.5) | 6.4 (1.3)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis on log-transformed HbA1c comparing the average HbA1c between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.985, Mixed Models Analysis; Difference in average HbA1c at 12 months between control and intervention groups; Mean percent change in HbA1c = 0.02, 95% CI 2-sided [-2.57 to 2.69] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

9. Secondary Outcome: Short Form (SF)-12 Mental Component Score (MCS)
Description: The SF-12 is a health-related quality of life measure that assesses general physical (PCS) and mental health (MCS) functioning and well-being, with the MCS score assessing mental health status. The investigators scored the SF-12 using QualityMetric's scoring software. MCS scores range from 0-100 with higher scores indicating better general menal health.
Time Frame: 12 months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 191 | 219
score on a scale | 47.2 (12.4) | 48.1 (11.4)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average 12-month MCS between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.806, Mixed Models Analysis; Difference in average SF-12 MCS score at 12 months between control and intervention groups; Mean Difference (Net) = -0.22, 95% CI 2-sided [-1.99 to 1.55] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

10. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: DBP values were obtained from the VA electronic health record. DBP is a measure of artery pressure when the heart rests between beats.
Time Frame: DBP closest to 12 months from baseline between 9-15 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 205 | 194
millimeters of mercury (mmHg) | 77.4 (8.0) | 77.2 (7.2)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average 12-month DBP between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.620, Mixed Models Analysis; Difference in average DBP at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.77 to 1.05] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

11. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: SBP values were obtained from the VA electronic health record. SBP is a measure of how much pressure blood is exerting against artery walls when the heart beats.
Time Frame: SBP closest to 12 months from baseline between 9-15 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
Number analyzed (Participants) | 205 | 194
millimeters of mercury (mmHg) | 127.3 (11.6) | 126.9 (13.3)
Statistical Analysis 1: Comparison: Behavioral Lifestyle Intervention vs Usual Care Control; Linear mixed model analysis comparing the average SBP between control and intervention groups. Our analysis controlled for randomization strata: age (less than or greater than/equal to 65), BMI (at least 30/less than 35, at least 35/less than 40, or at least 40/less than for 45), and population density (rural or urban), while random effects were used to account for within-person variability; Test type: Superiority; p = 0.987, Mixed Models Analysis; Difference in average SPB at 12 months between control and intervention groups; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-2.32 to 2.28] — Standard errors estimated using Kenward-Rogers adjustment for the denominator degrees of freedom

ADVERSE EVENTS:
Time Frame: We systematically collected adverse events (AE) by body system as part of the the 12- and 24-month follow-up survey process. For conditions that participants indicated were new since their baseline visit, study staff conducted electronic health record chart review for details of that condition.
Description: Adverse Events were monitored/assessed without regard to specific Adverse Event Terms.
Arm/Group | Behavioral Lifestyle Intervention | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 4/254 | 1/257
Serious Adverse Events (participants affected / at risk) | 47/254 | 42/257
Other Adverse Events (participants affected / at risk) | 124/254 | 105/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Lifestyle Intervention (N=254) | Usual Care Control (N=257)
Cardiovascular (Cardiac disorders) | 12 (16) | 18 (18)
Dermatological (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Gastrointestinal (Gastrointestinal disorders) | 10 (11) | 5 (5)
Hematological (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Metabolic (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Neurological (Nervous system disorders) | 4 (5) | 4 (4)
Psychological (Psychiatric disorders) | 3 (3) | 2 (2)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (7)
Renal/Urologic (Renal and urinary disorders) | 5 (5) | 3 (3)
Hepatobiliary (Hepatobiliary disorders) | 2 (2) | 1 (1)
Other (General disorders) | 11 (11) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Lifestyle Intervention (N=254) | Usual Care Control (N=257)
Cardiovascular (Cardiac disorders) | 7 (7) | 14 (15)
Dermatological (Skin and subcutaneous tissue disorders) | 19 (25) | 12 (13)
Gastrointestinal (Gastrointestinal disorders) | 21 (22) | 16 (16)
Hematological (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Metabolic (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 65 (79) | 38 (44)
Neurological (Nervous system disorders) | 18 (20) | 11 (11)
Psychological (Psychiatric disorders) | 5 (5) | 6 (6)
Pulmonary/Respiratory (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 16 (18)
Renal/Urologic (Renal and urinary disorders) | 11 (12) | 9 (11)
Hepatobiliary (Hepatobiliary disorders) | 1 (1) | 1 (1)
Other (General disorders) | 29 (33) | 22 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT03260140/Prot_SAP_000.pdf